CLINICAL TRIAL: NCT03467399
Title: Clinical Evaluation of a Cochlear Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5620
Record Dates: First submitted 2016-09-16; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear implant users (Experimental): This is a within-subject, repeated measures study. There was one arm in this study, each subject served as their own control. All subjects received all interventions.
  Interventions: Device: Nucleus 7 Cochlear Implant System

INTERVENTIONS:
Device: Nucleus 7 Cochlear Implant System — A new cochlear implant sound processor system.

SUMMARY:
The primary objective of this study is to assess the usability of a Cochlear implant system.

DETAILED DESCRIPTION:
Measure participant ratings on satisfaction of a Cochlear implant system via use of validated and non-validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older
2. At least 6 months experience with a Nucleus 24 series or later implant in at least one implanted ear
3. At least 3 months experience with the CP810,CP920 or CP910 sound processor
4. Fluent speaker in the language used to assess speech perception performance
5. Willingness to participate in and to comply with all requirements of the protocol
6. Able to score 30% or more at +15 SNR with CI alone on a sentence in babble test

Exclusion Criteria:

1. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device
2. Additional disabilities that would prevent participation in evaluations
3. Nucleus 22 Implant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Cochlear implant subjects' ratings on hearing performance, connectivity, streaming, phone use, comfort, retention, ease of use and controls obtained with their own Sound Processor and the CP1000 Sound Processor. | One year
  Non-inferiority of subjects' overall satisfaction ratings for the CP1000 Sound Processor and related components measured following 3 months of use, compared to subjects' overall satisfaction rating for their own Sound Processor and related components measured at study onset.

SECONDARY OUTCOMES:
Speech perception performance of the CP1000 Sound Processor in quiet and in noise. | One year
  Data to substantiate the speech perception scores of the subjects for different quiet and noise conditions for different configurations of sound processor and / or accessories.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brinson, Principal Investigator — Cochlear Ltd
Locations (1):
- Cochlear Ltd, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No